CLINICAL TRIAL: NCT05925881
Title: Arthroscopic Assisted Lower Trapezius Tendon Transfer vs Bridging Repair for Irreparable Rotator Cuff Tears: A Randomized Controlled Trial
Brief Title: Lower Trapezius Transfer vs Bridging Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ivan Wong, MD, MD, FRCS(C), Prinicipal Investigator, Professor, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52466
Record Dates: First submitted 2023-06-13; First posted 2023-06-29 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower Trapezius Tendon Transfer (Active Comparator): The lower trapezius tendon transfer arm will consist of patients randomized to this surgical procedure. This is an arthroscopically assisted open procedure that involves harvesting of the lower trapezius muscle tendon and re-grafting it onto to shoulder to repair massive rotator cuff tears.
  Interventions: Procedure: Surgical Repair of Large to Massive Rotator Cuff Tears
- Bridging Reconstruction Repair (Active Comparator): The bridging reconstruction repair arm will consist of patients randomized to this surgical procedure. This operation is arthroscopic, and involves the insertion of a human dermal allograft to the rotator cuff, sutured and anchored in a "bridging" fashion to repair massive rotator cuff tears.
  Interventions: Procedure: Surgical Repair of Large to Massive Rotator Cuff Tears

INTERVENTIONS:
Procedure: Surgical Repair of Large to Massive Rotator Cuff Tears — Surgical procedure to reconstruct the rotator cuff

SUMMARY:
The goal of this clinical trial is to compare the bridging reconstruction technique vs the lower trapezius tendon transfer in patients with massive irreparable rotator cuff tears.

The main questions it aims to answer are:

* comparing the outcomes of the two surgical techniques (BRR with an acellular human dermal allograft implant vs Arthroscopic Assisted LTT Transfer) on the maintenance of the acromiohumeral distance
* compare the outcomes of strength, range of motion, and patient reported quality of life scores between the two techniques

Participants will be randomized into one of two surgical treatment groups (bridging reconstruction or lower trapezius tendon transfer) and followed for a minimum of two years to compare the outcomes between groups.

DETAILED DESCRIPTION:
Research Plan: A total of 60 patients will be enrolled in the study. In the pre-operative period, there will be no additional time requirements for the patient, except for the informed consent process for the study. Routine radiographs including an AP and Y view of the shoulder as well as a pre-operative MRI are obtained for all patients undergoing rotator cuff surgery.

The patients will complete a structured clinical examination conducted by a sports medicine fellowship trained orthopaedic consultant. The examination will consist of range of motion testing by goniometer, range of motion testing evaluated by one's reach envelope, as well as strength testing by hand dynamometer. The patient will also complete the Western Ontario Rotator Cuff Index (WORC) questionnaire.

Randomization: Randomization will be done with a computer random number generator. Treatment conditions will be inserted in ordered opaque envelopes. Two groups (bridging reconstruction, and lower trapezius transfer) will be selected with 30 subjects each group.

Surgical Procedures: Wong et al. (2021) described the surgical procedure for patients in the "Bridging" group. The bursa will be debrided thoroughly, and rotator cuff edges will be shaved down to stable tissue. Following this, an acellular human dermal patch will be rehydrated in saline solution for 15 minutes. The patch is stretched to remove the manufacturing surface irregularities. The patch is then sewn in place with braided polyester suture material. Multiple sutures, approximately 5 to 10 mm apart from one another will be used. The medial sutures are placed into the remnants of supraspinatus and infraspinatus tendons. The patch is then attached to the greater tuberosity in a double row configuration.

The lower trapezius transfer will be performed as described by Wagner et. al. (2018). Patients will be placed in beach chair position, with the ipsilateral half of the back uncovered for surgical access. A 5-cm vertical skin incision will be made 1 cm from the medial border of scapula by the upper and lower edge of the lower trapezius tendon. The fat area at the inferior edge of the lower trapezius tendon will be identified, and the lower trapezius tendon will be completely released from spine of scapula and medially through opening of the superficial fascia. Two sutures in a Krakow configuration will be placed in the lower trapezius tendon. 2 sutures of different colors will be placed in the thick part of the allograft in a Krakow configuration. Designated ventral and dorsal aspects of the allograft will be marked. The infraspinatus fascia will be opened at the level of the medial incision. The sutures in the thick part of the allograft are then clamped to bring the graft intra-articular. Each of the Krakow sutures placed in the thick end of the allograft are passed to each of the 2 loadable suture anchors to attach the most distal part of the allograft, fixating the graft.

Postoperative protocol: The shoulder will be immobilized in a sling for one week postoperatively, and only passive forward flexion and external rotation will be allowed for eight weeks. The patient then progresses to active shoulder motion. Strengthening will begin at twelve weeks postoperatively. The patient will follow-up with the attending surgeon (IW) at 2 weeks post-operatively for a wound check. Then further clinical follow-up appointments will be at 6 weeks, 3 months, 6 months, 12 and 24 months, as per current clinical practice.

At the 6, 12, and 24 month visits the patient will again undergo the structured clinical examination conducted by a sports medicine fellowship trained orthopaedic consultant who is blinded to the patients' treatment group. The patient will also complete the WORC questionnaire at these follow-up appointments. Radiographs will be taken also to obtain the postoperative measurements. MRI will be done to assess healing at 12 months.

Analysis of Data: The data collected will be analyzed through SPSS version 24. Two-tailed independent t-tests will be performed for the WORC, acromiohumeral distance, range of motion, and strength measures comparing the two groups at most recent postoperative measurement. Repeated-measures ANOVA will be used to assess differences in WORC scores, range of motion and strength within each group between time points.

ELIGIBILITY:
Inclusion Criteria:

* magnetic resonance imaging (MRI) proven diagnosis of a massive rotator cuff tear
* tear size >5cm
* two-tendon, irreparable tear
* competent adult (>18 years of age)
* <50% muscle atrophy.

Exclusion Criteria:

* irreparable subscapular tear
* glenohumeral osteoarthritis
* WORC score > 70
* uncontrolled diabetes (Hgb A1C >7%)
* pregnancy
* presence of local or systemic infection
* inability to cooperate with and/or comprehend post-operative instructions
* cancer
* paralysis of the shoulder
* contracture of the shoulder
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Acromiohumeral Distance | 1 year
  The acromiohumeral distance is the shortest distance between the inferior aspect of the acromion to the closest part of the humeral head. This outcome will be measured by a single blinded assessor who has medical training (sports medicine trained surgical fellow). Acromiohumeral distance will be measured on MRI scans taken at one year post-op.

SECONDARY OUTCOMES:
Range of Motion | 1 year
  Range of motion will be measured by a single independent blinded assessor who has appropriate training (sports medicine trained surgical fellow). Range of motion will be assessed for forward flexion, abduction, internal rotation and external rotation. All measures will be conducted using a goniometer and recorded in degrees.
Strength | 1 year
  Strength will be measured by a single independent blinded assessor who has appropriate training (sports medicine trained surgical fellow). Strength will be measured during forward flexion, abduction of the shoulder, internal rotation and external rotation. All measures will be conducted using a handheld dynamometer and recorded in pounds.
Patient-reported Outcomes (PROs) | 1 year
  PROs will be measured using the Western Ontario Rotator Cuff Index (WORC) and the Disabilities of the Arm, Shoulder, and Hands Questionnaire (DASH). The WORC is a series of questions regarding patient quality of life and activities of daily living with a rotator cuff pathology. The score is a numerical value on a scale from 1-100, with lower values indicating better outcomes. WORC outcome scores will be calculated as the change in pre- to post-operative WORC, where a change in score greater than 11.7 points meets the minimum clinically important difference. The DASH is a 30-item, self-report questionnaire that measures physical function and symptoms in people with disorders of the upper limb/s. The score is a numerical value on a scale from 1-100, with lower values indicating better outcomes. DASH outcome scores will compare the pre- to post-operative DASH, with a change in score greater than 10.81 indicating the minimum clinically important difference has been met.

CONTACTS AND LOCATIONS:
Locations (1):
- 5955 Veterans' Memorial Lane Room 2106, VMB, Halifax, Nova Scotia, Canada